CLINICAL TRIAL: NCT02552134
Title: HEPA Steiermark: Standardised Regional Sport-club Based Exercise Programmes
Brief Title: Standardised Regional Sport-club Based Exercise Programmes
Acronym: SRS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sportunion Österreich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SPU HEPA
Record Dates: First submitted 2015-09-15; First posted 2015-09-16 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-09

CONDITIONS: Physical Activity
Keywords: Access to physical activity resources, community based exercise programme, sports-clubs, health resort,
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- frequent participation (Experimental): After termination of a stationary stay in a health resort, participants will visit an initial standardised regional sport club based exercise programme for 12 sessions at the place of the residence.
  Interventions: Other: exercise training
- medium participation (Experimental): After termination of a stationary stay in a health resort, participants will visit an initial standardised regional sport club based exercise programme for 12 sessions at the place of the residence
  Interventions: Other: exercise training
- low participation (Experimental): After termination of a stationary stay in a health resort, participants will visit an initial standardised regional sport club based exercise programme for 12 sessions at the place of the residence
  Interventions: Other: exercise training
- recommendation to be active (Active Comparator): During the stay in the health care resort participants are introduced to be active in the future. They will receive a brochure "Physical Activity: Health for all".
  Interventions: Other: recommendation to be active

INTERVENTIONS:
Other: exercise training
  Arms: frequent participation; low participation; medium participation
Other: recommendation to be active
  Arms: recommendation to be active

SUMMARY:
Background: More than 10% of the adult population in Styria, a federal state in the south of Austria, is allotted to a stationary stay at a health resort each year. In practice approximately 50.000 adults receive these stays that are financed from the health insurance companies and that last up to 3 weeks. The target group for theses stays is the general population aged between 30 and 65 years that shows minor health deficits like back pain or risk factors for cardio-metabolic diseases. The treatment during the stays consists of exercise, nutritional and psychological interventions. Thus the increase of physical activity is an important goal that is focussed during the stationary stay. Because of the absence of regional facilities that are linked to the resorts and that provide accesses to standardised regional programmes sustainability is questionable.

Methods/Design: This prospective controlled open label study compares two study groups. After a stationary stay at a health resort patient are allocated to a standardised, regional sports-club based exercise programme or to another group, where only written hand-outs are provided. The primary outcome is the weekly level of health enhancing physical activity which is objectively measured with an accelerometer and an activity log-book. Additionally, social determinants are requested, fitness and anthropometric measurements are done at baseline until 12 months. Beside the changes in measurable parameters, processes are evaluated accurately. Consequently the gateway - function of the health resort is analysed.

Discussion: The structured cooperation between the health sector, where health resorts informing and assigning patients to regional sports-clubs and the sports sector potentially provides a wide network of standardised programmes. Within this study we aim to evaluate the sustainability of stationary stays and a continuing regional standardised exercise programme.

ELIGIBILITY:
Inclusion Criteria:

* Austrian physical activity recommendations for substantial health benefits are not reached. (Weekly < 150 Minutes of aerobic moderate intense physical activity, or < 75 minutes of aerobic vigorous intense physical activity or an equal combination as well as and/or muscle-strengthening activities at least twice a week are not realised.)
* Stationary stay at a health resort
* Physical activity in the patient's responsibility is recommended
* Systolic blood pressure at rest ≤ 90 mm/Hg
* Diastolic blood pressure at rest ≤ 140 mm/Hg

Exclusion Criteria:

* More than 10% planned or unplanned weight loss / weight gain during the last 6 months
* Pregnancy
* Indication for stationary or outpatient rehabilitation based on the
* Untreated coronary heart disease
* Untreated micro- or macrovascular artery disease

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-03 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
the weekly level of accelerometer determined health enhancing physical activity, measured as minutes of moderate and vigorous physical activity | 7 complete consecutive days

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Titze, Dr, Study Chair — Institut für Sportwissenschaften der Karl-Franzens-Universität Graz
Locations (1):
- University of Graz, Graz, Styria, Austria

REFERENCES:
- [Derived] Lackinger C, Strehn A, Dorner TE, Niebauer J, Titze S. Health resorts as gateways for regional, standardised, sports club based exercise programmes to increase the weekly time of moderate- to vigorous-intensity physical activity: study protocol. BMC Public Health. 2015 Dec 21;15:1265. doi: 10.1186/s12889-015-2581-9. PMID 26692015